CLINICAL TRIAL: NCT06926569
Title: Single High-dose of Liposomal Amphotericin B in Combination With B/F/TAF for HIV/AIDS-associated Talaromycosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Yinzhong Shen, Principal Investigator, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GKT1200; IN-US-131-7590 (Other Grant/Funding Number: Gilead Sciences, Inc)
Record Dates: First submitted 2025-03-21; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: HIV/AIDS-associated Talaromycosis
Keywords: HIV/AIDS-associated talaromycosis
MeSH Terms: interventions — Amphotericin B; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single high-dose L-AmB group (Experimental): After enrollment, participants will be 1:1 randomly assigned into two groups for induction therapy after informed consent: single high-dose L-AmB group (10 mg/kg single intravenous dose of L-AMB) and control group (amphotericin B deoxycholate(AmBD) at 0.5-0.7 mg/kg/d intravenously for 14 days as the standard of care recommended by local guidelines).Thereafter, all participants in both groups will start consolidation therapy within 24 hours of the induction treatment, 200mg itraconazole(or voriconazole) q12h will be given for 10 weeks. After consolidation therapy, all participants will take oral itraconazole 200mg qd as secondary prophylaxis until their CD4+ cell counts are higher than 100cells/mm3 for at least 6 months. For the antiretroviral therapy, all participants will start B/F/TAF qd within 7 days after initiating antifungal therapy.
  Interventions: Drug: AmBisome
- Control group (Other): After enrollment, participants will be 1:1 randomly assigned into two groups for induction therapy after informed consent: single high-dose L-AmB group (10 mg/kg single intravenous dose of L-AMB) and control group (amphotericin B deoxycholate(AmBD) at 0.5-0.7 mg/kg/d intravenously for 14 days as the standard of care recommended by local guidelines).Thereafter, all participants in both groups will start consolidation therapy within 24 hours of the induction treatment, 200mg itraconazole(or voriconazole) q12h will be given for 10 weeks. After consolidation therapy, all participants will take oral itraconazole 200mg qd as secondary prophylaxis until their CD4+ cell counts are higher than 100cells/mm3 for at least 6 months. For the antiretroviral therapy, all participants will start B/F/TAF qd within 7 days after initiating antifungal therapy.
  Interventions: Drug: Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B — After enrollment, participants will be 1:1 randomly assigned into two groups for induction therapy after informed consent: single high-dose L-AmB group (10 mg/kg single intravenous dose of L-AMB) and control group (amphotericin B deoxycholate(AmBD) at 0.5-0.7 mg/kg/d intravenously for 14 days as the standard of care recommended by local guidelines).Thereafter, all participants in both groups will start consolidation therapy within 24 hours of the induction treatment, 200mg itraconazole(or voriconazole) q12h will be given for 10 weeks. After consolidation therapy, all participants will take oral itraconazole 200mg qd as secondary prophylaxis until their CD4+ cell counts are higher than 100cells/mm3 for at least 6 months. For the antiretroviral therapy, all participants will start B/F/TAF qd within 7 days after initiating antifungal therapy
  Arms: Control group
Drug: AmBisome — After enrollment, participants will be 1:1 randomly assigned into two groups for induction therapy after informed consent: single high-dose L-AmB group (10 mg/kg single intravenous dose of L-AMB) and control group (amphotericin B deoxycholate(AmBD) at 0.5-0.7 mg/kg/d intravenously for 14 days as the standard of care recommended by local guidelines).Thereafter, all participants in both groups will start consolidation therapy within 24 hours of the induction treatment, 200mg itraconazole(or voriconazole) q12h will be given for 10 weeks. After consolidation therapy, all participants will take oral itraconazole 200mg qd as secondary prophylaxis until their CD4+ cell counts are higher than 100cells/mm3 for at least 6 months. For the antiretroviral therapy, all participants will start B/F/TAF qd within 7 days after initiating antifungal therapy.
  Arms: Single high-dose L-AmB group

SUMMARY:
This study aims to compare the efficacy and safety of a single high-dose Liposomal Amphotericin B (L-AMB) against conventional Amphotericin B deoxycholate (AmBD) for HIV-associated Talaromycosis.

The investigators hypothesize that L-AMB induction therapy (10 mg/kg) is non-inferior to AmBD (0.5-0.7 mg/kg/d) in efficacy and has an improved safety profile.

The study's primary objective is to provide evidence supporting the guideline recommendation of single high-dose L-AMB for HIV-infected individuals with talaromycosis, while validating L-AMB's efficacy and safety in China.

Study Design: Multi-center, randomized controlled trial comparing single high-dose L-AMB to guideline-recommended AmBD induction therapy for HIV-associated talaromycosis. Participants are HIV-infected adults (≥18 years) with confirmed talaromycosis by microscopy or culture.

Interventions:

1. L-AMB group receives a single intravenous dose of 10 mg/kg L-AMB.
2. Control group receives intravenous AmBD at 0.5-0.7 mg/kg/d for 14 days.
3. Both groups start consolidation therapy with itraconazole 200mg q12h for 10 weeks within 24 hours post-induction.
4. Secondary prophylaxis with itraconazole 200mg qd until CD4+ cell counts exceed 100cells/mm³ for at least 6 months.
5. All start B/F/TAF qd within 7 days post-antifungal therapy.

Primary Objective： This multicenter study compares efficacy/safety of single high-dose L-AMB vs standard AmBD (2-week) induction for HIV-associated talaromycosis, generating evidence to support L-AMB guidelines in Chinese populations.

Secondary Objectives： Evaluate feasibility/safety of initiating B/F/TAF within 7 days post-antifungal therapy, providing evidence for rapid ART guidelines in these patients.

Endpoints:

* Primary: Proportion achieving clinical resolution on day 14.
* Secondary: Overall survival, renal function, anemia, liver function, adverse events grade 3 or higher on day 14; time to clinical resolution and sterile blood cultures; survival, HIV viral suppression, CD4+ T-cell counts, adverse events (including IRIS), ART persistency, and patient-reported outcomes at weeks 4, 12, and 24.

Sample Size: 58 participants per group (116 total), considering a 10% dropout rate.

DETAILED DESCRIPTION:
Scientific Basis/Rationale Talaromycosis caused by Talaromyces marneffei (TM) is a highly aggressive fungal infection predominantly observed in people living with HIV (PLWH). The mortality rate for untreated talaromycosis ranges from 75% to 97%, and where the infection is uncontrolled in PLWH, the fatality rate can approach 100%. Talaromycosis is endemic in South-East Asia and parts of China and India, contributing to a significant burden in these areas [1]. Notebly, talaromycosis is responsible for one-sixth of AIDS-related hospitalizations and exhibits a high mortality rate. In China, approximately 99% of TM infections are concentrated in the southern region, where it is one of the leading causes of AIDS-associated deaths. The endemic range of talaromycosis has expanded beyond traditional regions in southern China, Southeast Asian countries and Northeast India, now encompassing 34 countries and regions worldwide. The case fatality rate for untreated talaromycosis remains alarmingly high, between 75% and 100% [1, 2].

The antifungal management of talaromycosis in PLWH involves three phases: induction, consolidation and maintenance, with the induction phase being of paramount importance. Based on findings from the Itraconazole versus AmphotericinB for Penicilliosis (IVAP) studies and observational studies, the DHHS guidelines recommend amphotericin B for induction therapy, with liposomal amphotericin B (L-AMB) as the preferred agent due to its superior safety profile and favorable clinical outcome [3]. Historically, Chinese AIDS treatment guidelines have recommended amphotericin B deoxycholate (AMB d, 0.5-0.7mg/kg/d) as the standard therapy for AIDS-associated talaromycosis. However, the nephrotoxicity and adverse effects including anemia and electrolyte disturbances associated with AMB d have resulted in suboptimal therapeutic outcomes [4, 5]. L-AMB has demonstrated reduced toxicity, enhanced safety and prolonged tissue half-life [2, 6]. Following its introduction to China in June 2023, L-AMB (3-5mg/kg/d) is now recommended in updated local guidelines for HIV-associated talaromycosis [7]. Nevertheless, given the relatively recent clinical availability of L-AMB, clinical experience and data on its use in people living with HIV (PLWH) in China remain limited.

The use of single high-dose L-AMB has been explored in clinical trials for various fungal infections [8, 9]. Due to its reduced drug-induced toxicity, higher doses of L-AMB can be administered safely [10]. WHO has endorsed single high-dose L-AMB for the treatment of cryptococcal meningitis based on findings from the Ambition study [10]. Additionally, a Phase II trial investigating HIV/AIDS-associated disseminated histoplasmosis showed that a one-day induction therapy with 10 mg/kg L-AMB was both safe and effective [6]. Despite these promising findings, this therapeutic approach has not yet been rigorously evaluated in the context of HIV-associated talaromycosis.

The optimal timing of initiation of antiretroviral therapy (ART) for HIV-associated talaromycosis remains uncertain. DHHS guidelines recommend starting ART 1 week after initiating amphotericin B therapy [3]. Bictegravir/Emtricitabine/Tenofovir Alafenamide Fumarate (B/F/TAF) is a single-tablet regimen recommended for the rapid initiation of ART (within 7 days after HIV diagnosis) in PLWH, offering potent viral suppression and a favorable safety profile. However, there is a paucity of data regarding the use of regimen in PLWH with advanced opportunistic infection (OIs), including HIV-associated talaromycosis.

Hypothesis The investigators hypothesize that a single high dose regimen of L-AMB (10 mg/kg) as induction therapy for HIV-associated talaromycosis is non-inferior to the conventional administration of AmBD (0.5-0.7mg/kg/d) in terms of efficacy and is associated with an improved safety profile. Specifically, the investigators expected that key clinical outcomes including the proportion of participants who achieve clinical resolution on day 14, the rate of fungal clearance during the induction phase, the time to clinical symptom remission, and the mortality rate of patients will be comparable to those observed with conventional AmBD therapy. Additionally, the investigators anticipant a reduction in the incidence of grade 3 or above adverse events, defined by clinical or laboratory criteria. Furthermore, the investigators propose that rapid initiation of B/F/TAF within 7 days after antifungal therapy is feasible in this population. This can be demonstrated by observing indicators such as HIV suppression rate, occurrence and progression of immune reconstitution inflammatory syndrome (IRIS), the absolute median or percentage change in laboratory values (such as CD4 T cell counts) as well as the patient-reported outcomes(PROs).

Primary Objective This prospective multicenter clinical study aims to compare the efficacy and safety of a single high-dose L-AMB with guidelines-recommended first-line induction therapy (2 weeks of AmBD) for the treatment of HIV-associated talaromycosis. The study seeks to provide robust, high-quality evidence to support the guideline recommendation of a single high dose of L-AMB for HIV-infected individuals with talaromycosis, while validating and accumulating efficacy and safety data of L-AMB in the Chinese population.

Secondary Objectives The secondary objectives include assessing the feasibility of rapid initiation of B/F/TAF within 7 days after antifungal therapy initiation. The study aims to provide high-quality evidence to support guideline recommendations on the rapid initiation of B/F/TAF in HIV-associated talaromycosis patients, while verifying its safety and efficacy.

Study Design and Research Methods This is a multi-center randomized controlled trial. This trial intends to evaluate the efficacy and safety of single high-dose L-AMB for induction therapy for HIV-associated talaromycosis, in comparison to amphotericin B deoxycholate (AmBD) as recommended by the local guidelines.

Eligible participants were HIV-infected adults (18 years of age) who had talaromycosis that was confirmed by either microscopy or culture. Participants will be recruited based on predefined inclusion and exclusion criteria. After enrollment, participants will be 1:1 randomly assigned into two groups for induction therapy after informed consent: single high-dose L-AmB group (10 mg/kg single intravenous dose of L-AMB) and control group (amphotericin B deoxycholate(AmBD) at 0.5-0.7 mg/kg/d intravenously for 14 days as the standard of care recommended by local guidelines).Thereafter, all participants in both groups will start consolidation therapy within 24 hours of the induction treatment, 200mg itraconazole(or voriconazole) q12h will be given for 10 weeks. After consolidation therapy, all participants will take oral itraconazole 200mg qd as secondary prophylaxis until their CD4+ cell counts are higher than 100cells/mm3 for at least 6 months. For the antiretroviral therapy, all participants will start B/F/TAF qd within 7 days after initiating antifungal therapy.

All participants will be hospitalized during the initial 2-week period of the trial, during which time administration of therapy is directly observed. Patients will be closely monitored during the first 2-week inpatient period and then followed up in outpatient clinics for 6 months. The primary endpoint is the proportion of participants who achieve clinical resolution on day 14, defined as resolution of symptoms/signs attributable to talaromycosis, such as fever and rash (temperature below 38 for more than 3 days, improvement of rash) and sterile blood cultures, except for manifestations that are expected to last for more than 14 days after treatment initiation: hepatosplenomegaly, jaundice and pancytopenia. Secondary endpoints are also determined on day 14 and included overall survival, renal function abnormalities, anemia, and liver function abnormalities and clinical or laboratory-defined adverse events of grade 3 or higher. Overall survival, HIV viral suppression, CD4+ T-cell counts, adverse events (including immune reconstitution inflammatory syndrome, IRIS), ART persistency and patient-reported outcomes will also be evaluated at week 4, 12 and 24.

Each group consists of 58 participants(116 in total). Subjects will be recruited at four clinical centers in southern China, with preliminary allocations as follows: Shanghai Public Health Clinical Center (22 cases) , Chest Hospital of Guangxi Zhuang Autonomous Region(43 cases), Fujian Mengchao Hepatobiliary Hospital (20 cases), and Guiyang Public Health Center (31 cases).

Number of Sites 4

Treatment Regimen

1. Regimen, dosage and usage of anti-talaromycosis therapeutic drugs:

   Experimental group(Single high-dose L-AmB group): 10 mg/kg single intravenous dose of L-AMB Control group: amphotericin B deoxycholate(AmBD) at 0.5-0.7 mg/kg/d intravenously for 14 days Within 24h after induction treatment, all participants will start 200mg itraconazole(or voriconazole) q12h for 10 weeks for consolidation therapy. Thereafter, itraconazole 200mg qd as secondary prophylaxis until their CD4+ cell counts are higher than 100cells/mm3 for at least 6 months.
2. Regimen, dosage and usage of antiretroviral therapy: Bictegravir/Emtricitabine/Tenofovir Alafenamide Fumarate (BIC/FTC/TAF: 50 mg/200 mg/25 mg, qd oral) for participants in both groups
3. Timing of antiretroviral therapy: all participants will initiate B/F/TAF within 1 week after initiation of antifungal therapy

Inclusion Criteria

1. Aged 18 and above
2. ART naive
3. HIV positive individuals
4. Confirmed Talaromycosis diagnosed by culture/microscopy

Exclusion Criteria

1. Pregnancy or lactating women;
2. Central nervous system involvement (assessed either through clinical manifestations or cerebrospinal fluid analysis);
3. Known allergy to AMB d/L-AMB, or the concomitant use of medications known to interact with AMB d/L-AMB;
4. Alanine aminotransferase or aspartate aminotransferase levels exceeding 400 U/L;
5. Absolute neutrophil count below 500/mm3;
6. Creatinine clearance below 30 mL/min (calculated using the Cockcroft and Gault equation);
7. Concurrent diagnosis of cryptococcal meningitis;
8. Concurrent treatment with rifampicin;
9. Previous treatment for talaromycosis lasting more than 48 hours.

Primary Endpoint The primary endpoint is the proportion of participants who achieve clinical resolution on day 14 .

Clinical resolution defined as resolution of symptoms/signs attributable to talaromycosis, such as fever and rash (temperature below 38 for more than 3 days, improvement of rash) and sterile blood cultures, except for manifestations that are expected to last for more than 14 days after treatment initiation: hepatosplenomegaly, jaundice and pancytopenia [11].

Secondary Endpoint The secondary endpoints are: 1. overall survival, renal function abnormalities, anemia, and liver function abnormalities and clinical or laboratory-defined adverse events of grade 3 or higher on d14; 2.the time to clinical resolution, defined as resolution of symptoms/signs attributable to talaromycosis, such as fever and rash (temperature below 38 for more than 3 days, improvement of rash) and sterile blood cultures, except for manifestations that are expected to last for more than 14 days after treatment initiation; 3. the time to achieve sterile blood cultures, the rate of fungal clearance from blood at 7 and14 days over the course of induction therapy; 4. overall survival, HIV viral suppression, CD4+ T-cell counts, adverse events (including immune reconstitution inflammatory syndrome, IRIS), ART persistency and patient-reported outcomes at week 4, 12 and 24.

Sample Size Justification/Statistical Analysis Using a non-inferiority design, assuming an expected proportion of favorable response equals to 95% [11], a sample size of 52 subjects per arm would provide the trial with 80% of power to show non-inferiority of the alternative arms to the local guideline recommended regimen, given a specified non-inferiority margin of 12% and 1-side = 0.025. Considering a dropout rate of 10%, the sample size per arm was calculated to 58 patients, and the total sample size for the study was 116 patients. Statistical software SAS 9.4 or above will be used for analysis in this study. Comparisons between groups of classified data will be made using Chi-square test or fisher exact probability method; Comparison between two sets of continuous data will be performed using Wilcoxon rank sum test or T test. Statistical tests will be two-sided tests with a significance level of 0.05 if not otherwise specified.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and above
2. ART naive
3. HIV positive individuals
4. Confirmed Talaromycosis diagnosed by culture/microscopy

Exclusion Criteria:

1. Pregnancy or lactating women;
2. Central nervous system involvement (assessed either through clinical manifestations or cerebrospinal fluid analysis);
3. Known allergy to AMB d/L-AMB, or the concomitant use of medications known to interact with AMB d/L-AMB;
4. Alanine aminotransferase or aspartate aminotransferase levels exceeding 400 U/L;
5. Absolute neutrophil count below 500/mm3;
6. Creatinine clearance below 30 mL/min (calculated using the Cockcroft and Gault equation);
7. Concurrent diagnosis of cryptococcal meningitis;
8. Concurrent treatment with rifampicin;
9. Previous treatment for talaromycosis lasting more than 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
the proportion of participants who achieve clinical resolution on day 14 | 14 days
  The primary endpoint is the proportion of participants who achieve clinical resolution on day 14 .
  Clinical resolution defined as resolution of symptoms/signs attributable to talaromycosis, such as fever and rash (temperature below 38 for more than 3 days, improvement of rash) and sterile blood cultures, except for manifestations that are expected to last for more than 14 days after treatment initiation: hepatosplenomegaly, jaundice and pancytopenia.

SECONDARY OUTCOMES:
Overall Survival | 14 days
  overall survival one day14
Adverse Events | 14 days
  renal function abnormalities, anemia, and liver function abnormalities and clinical or laboratory-defined adverse events of grade 3 or higher on d14.
The Time to Clinical Resolution | one year
  defined as resolution of symptoms/signs attributable to talaromycosis, such as fever and rash (temperature below 38 for more than 3 days, improvement of rash) and sterile blood cultures, except for manifestations that are expected to last for more than 14 days after treatment initiation
The Time to Achieve Sterile Blood Cultures | 14 days
  the rate of fungal clearance from blood at 7 and14 days over the course of induction therapy
HIV viral suppression | 24 weeks
  HIV viral suppression at week 4, 12 and 24
CD4+ T-cell counts | 24 weeks
  CD4+ T-cell counts at week 4, 12 and 24
ART persistency | 24 weeks
  ART persistency at week 4, 12 and 24
Patient-reported Outcomes | 24 weeks
  patient-reported outcomes at week 4, 12 and 24

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le T, Kinh NV, Cuc NTK, Tung NLN, Lam NT, Thuy PTT, Cuong DD, Phuc PTH, Vinh VH, Hanh DTH, Tam VV, Thanh NT, Thuy TP, Hang NT, Long HB, Nhan HT, Wertheim HFL, Merson L, Shikuma C, Day JN, Chau NVV, Farrar J, Thwaites G, Wolbers M; IVAP Investigators. A Trial of Itraconazole or Amphotericin B for HIV-Associated Talaromycosis. N Engl J Med. 2017 Jun 15;376(24):2329-2340. doi: 10.1056/NEJMoa1613306. PMID 28614691
- [Background] Adler-Moore J, Lewis RE, Bruggemann RJM, Rijnders BJA, Groll AH, Walsh TJ. Preclinical Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antifungal Activity of Liposomal Amphotericin B. Clin Infect Dis. 2019 May 2;68(Suppl 4):S244-S259. doi: 10.1093/cid/ciz064. PMID 31222254
- [Background] Sundar S, Chakravarty J, Agarwal D, Rai M, Murray HW. Single-dose liposomal amphotericin B for visceral leishmaniasis in India. N Engl J Med. 2010 Feb 11;362(6):504-12. doi: 10.1056/NEJMoa0903627. PMID 20147716
- [Background] Jarvis JN, Lawrence DS, Meya DB, Kagimu E, Kasibante J, Mpoza E, Rutakingirwa MK, Ssebambulidde K, Tugume L, Rhein J, Boulware DR, Mwandumba HC, Moyo M, Mzinganjira H, Kanyama C, Hosseinipour MC, Chawinga C, Meintjes G, Schutz C, Comins K, Singh A, Muzoora C, Jjunju S, Nuwagira E, Mosepele M, Leeme T, Siamisang K, Ndhlovu CE, Hlupeni A, Mutata C, van Widenfelt E, Chen T, Wang D, Hope W, Boyer-Chammard T, Loyse A, Molloy SF, Youssouf N, Lortholary O, Lalloo DG, Jaffar S, Harrison TS; Ambition Study Group. Single-Dose Liposomal Amphotericin B Treatment for Cryptococcal Meningitis. N Engl J Med. 2022 Mar 24;386(12):1109-1120. doi: 10.1056/NEJMoa2111904. PMID 35320642
- [Background] Chinese guidelines for diagnosis and treatment of human immunodeficiency virus infection/acquired immunodeficiency syndrome (2024 edition), 10.3760/cma.j.cn311365-20240328-00081.
- [Background] Pasqualotto AC, Lana DD, Godoy CSM, Leitao TDMJS, Bay MB, Damasceno LS, Soares RBA, Kist R, Silva LR, Wiltgen D, Melo M, Guimaraes TF, Guimaraes MR, Vechi HT, de Mesquita JRL, Monteiro GRG, Adenis A, Bahr NC, Spec A, Boulware DR, Israelski D, Chiller T, Falci DR. Single High Dose of Liposomal Amphotericin B in Human Immunodeficiency Virus/AIDS-Related Disseminated Histoplasmosis: A Randomized Trial. Clin Infect Dis. 2023 Oct 13;77(8):1126-1132. doi: 10.1093/cid/ciad313. PMID 37232940
- [Background] Bicanic T, Bottomley C, Loyse A, Brouwer AE, Muzoora C, Taseera K, Jackson A, Phulusa J, Hosseinipour MC, van der Horst C, Limmathurotsakul D, White NJ, Wilson D, Wood R, Meintjes G, Harrison TS, Jarvis JN. Toxicity of Amphotericin B Deoxycholate-Based Induction Therapy in Patients with HIV-Associated Cryptococcal Meningitis. Antimicrob Agents Chemother. 2015 Dec;59(12):7224-31. doi: 10.1128/AAC.01698-15. Epub 2015 Sep 8. PMID 26349818
- [Background] Ullmann AJ. Nephrotoxicity in the setting of invasive fungal diseases. Mycoses. 2008;51 Suppl 1:25-30. doi: 10.1111/j.1439-0507.2008.01525.x. PMID 18471158
- [Background] Panel on Guidelines for the Prevention and Treatment of Opportunistic Infections in Adults and Adolescents with HIV. Guidelines for the Prevention and Treatment of Opportunistic Infections in Adults and Adolescents with HIV. National Institutes of Health, Centers for Disease Control and Prevention, HIV Medicine Association, and Infectious Diseases Society of America. Available at https://clinicalinfo.hiv.gov/en/guidelines/adult-andadolescent-opportunistic-infection. Accessed 25/6/2024
- [Background] Wang F, Han R, Chen S. An Overlooked and Underrated Endemic Mycosis-Talaromycosis and the Pathogenic Fungus Talaromyces marneffei. Clin Microbiol Rev. 2023 Mar 23;36(1):e0005122. doi: 10.1128/cmr.00051-22. Epub 2023 Jan 17. PMID 36648228
- [Background] Guo P, Li L, Tang X. Advances in diagnosis and treatment of talaromycosis in patients with AIDS. Chin Med J (Engl). 2022 Nov 20;135(22):2687-2689. doi: 10.1097/CM9.0000000000002506. No abstract available. PMID 36719357
- [Derived] Yan X, Meng X, Song W, Liu L, Chen J, Zhang R, Shen Y. Single high-dose liposomal amphotericin B plus B/F/TAF for AIDS-associated talaromycosis in China: a multicentre randomised controlled trial protocol. BMJ Open. 2025 Nov 19;15(11):e105648. doi: 10.1136/bmjopen-2025-105648. PMID 41263912